CLINICAL TRIAL: NCT03588793
Title: The Reliability and Validity of Outcome Measures for People Who Have Phantom Limb Pain
Brief Title: Reliability and Validity of Outcome Measures for Phantom Limb Pain
Status: Completed | Type: Observational
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Andrew Graham, PhD candidate, Teesside University
Other Study IDs: TU243418
Record Dates: First submitted 2018-06-25; First posted 2018-07-17 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Phantom Limb Pain
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Two Point Discrimination — Validity of mechanism in phantom limb pain i.e. cortical reorganisation to be tested using comparison of data from interventions above
  Other Names: Implicit Motor Imagery Testing

SUMMARY:
Phantom limb pain (PLP) is experienced by 60-80% of all people who have had an amputation. This persistent pain condition can impact on independence, activities of daily living and overall quality of life.

While there is some research into PLP there is no consensus on appropriate outcome measures and there is (to our knowledge) neither guideline nor literature evidence on the reliability and validity of outcomes measures for this patient group. Such measures are vital to the robust evaluation of any interventions and/or monitoring progression.

The aim of the proposed study is to assess the reliability and validity of four self-report questionnaires (Visual Analog Scale (VAS) for pain, Short Form McGill Pain Questionnaire 2 (SFMPQ-2), Trinity Amputation and Prosthetic Evaluation Scale (TAPES), a health-related quality of life measure (EQ-5D-L), a pain diary, a left/right limb judgement task (Implicit Motor Imagery Testing - IMIT) and the two-point discrimination (TPD)test.

The data will be collated and statistically analysed to assess how stable each of the measures are over time (intra session reliability) and how each measure co-relates with the others (validity).

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years At least six months post amputation (date of surgery) The amputation must be above wrist/ankle. Are currently experiencing PLP which has persisted for at least 3 months or more They rate their PLP as ≥3 on a 0-10 scale on at least 2 days in the preceding week Concomitant medications;

Exclusion Criteria:

* Participating in any research trial of any intervention hypothesised to affect PLP.

Currently under-going active prosthetic rehabilitation e.g. walking training sessions or upper limb rehabilitation sessions.

Any current non-prescribed substance dependency An inability to understand and follow basic instructions - both the two-point discrimination test and left/right limb judgement task requires the participant to follow basic/simple instructions.

Any person, otherwise eligible, who commences any treatment for PLP (physical or pharmacological, prescribed or non-prescribed) will be withdrawn from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Amputees
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Statistical analysis of change in Visual Analogue Scale (VAS) for pain scores | Administered on 2 separate occasions, 7-14 days apart
  Intra-rater reliability analysis

SECONDARY OUTCOMES:
Statistical analysis of change in EQ-5D-L scores | Administered on 2 separate occasions, 7-14 days apart
  Health related Quality of Life questionnaire. Intra-rater reliability analysis
Statistical analysis of change in Short Form McGill Pain Questionnaire 2 (SF-MPQ-2) scores | Administered on 2 separate occasions, 7-14 days apart
  Intra-rater reliability analysis
Statistical analysis of change in Trinity Amputation and Prosthetic Evaluation Score - Revised (TAPES-R) - Amended version to include phantom limb pain and demographics questions | Administered on 2 separate occasions, 7-14 days apart
  Intra-rater reliability

CONTACTS AND LOCATIONS:
Locations (1):
- Teesside University School of Health & Social Care, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided